CLINICAL TRIAL: NCT00456066
Title: Assessment of Efficacity of Coronary Thromboaspiration (Export System) Performed Before Angioplasty on Infarct Size in Patients Treated by Coronary Percutaneous Interventions During Acute Phase.
Brief Title: Coronary Thromboaspiration and Infarct Size
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Janusz LIPIECKI, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU63-0018
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Ischemic Heart Disease; Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Thromboaspiration; Infarct size; Left ventricular remodelling
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: Export Aspiration System — Patients scheduled for emergency angioplasty

SUMMARY:
Distal embolization can occur during coronary angioplasty performed in the acute phase of myocardial infarction and is associated with poor long-term outcome. We hypothesize that the use of a system allowing thrombus aspiration before angioplasty and stent implantation will limit infarct size and its severity.

DETAILED DESCRIPTION:
Patients scheduled for emergency angioplasty in the acute phase of a first ST-elevation myocardial infarction will be treated either by thromboaspiration followed by angioplasty or by angioplasty alone. The infarct size and severity will be assessed by ce-MRI and rest Tc99m-mibi gated SPECT performed during initial hospital stay (5th-8th day). A control MRI will be performed at 6-month follow-up to analyse the evolution of left ventricular volumes.

ELIGIBILITY:
Inclusion Criteria:

* acute phase of myocardial infarction (>48 hours from the onset of chest pain)
* stable hemodynamic conditions
* completely occluded infarct related artery

Exclusion Criteria:

* heart failure signs in the acute phase
* contra indication for MRI or SPECT IMAGING

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Infarct size and severity assessed by ce-MRI and rest Tc99m-mibi gated SPECT | by ce-MRI and rest Tc99m-mibi gated SPECT

SECONDARY OUTCOMES:
Probability of evolution toward left ventricular remodelling (defined as an increase of end-diastolic volume of>20% between the acute phase and 6-montcontrol) | of end-diastolic volumeof>20% between the acute phase and 6-montcontrol)

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Lipiecki, Pr, Principal Investigator
Locations (1):
- Departement of Cardiology and Radiology, University Hospital, and Departement of Nuclear Medicine, Jean Perrin Cancer Centre, Clermont-Ferrand, Auvergne, France